CLINICAL TRIAL: NCT03497780
Title: Longitudinal Assessment of Cartilage Injury and Remodeling After Anterior Cruciate Ligament Rupture and Reconstruction: A Correlational Study of Synovial Inflammation, Functional Imaging, Clinical Outcomes, and Cartilage Biomarkers
Brief Title: Longitudinal Assessment of Cartilage Injury and Remodeling After Anterior Cruciate Ligament Rupture and Reconstruction:
Status: Terminated | Type: Observational
Why Stopped: Due to staff departure, study is being discontinued per allocation of resources.
Sponsor: University of Michigan (Other)
Collaborators: Peking University Health Science Center (Other)
Responsible Party: Principal Investigator, Tristan Maerz, Research Investigator, University of Michigan
Other Study IDs: HUM00137279
Record Dates: First submitted 2018-03-23; First posted 2018-04-13 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture; ACL Injury; Healthy
Keywords: Healthy Volunteers; ACL (Anterior Cruciate Ligament) tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Lacerations | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ACL Tear: Patients with ACL tears
  Interventions: Procedure: Anterior cruciate ligament reconstruction
- Healthy Subjects: Healthy subjects

INTERVENTIONS:
Procedure: Anterior cruciate ligament reconstruction — Primary surgical reconstruction of the rupture anterior cruciate ligament
  Groups: ACL Tear

SUMMARY:
The proposed study will establish novel relationships between intra-articular mesenchymal stem cell (MSC) recruitment, synovial inflammation, biomarkers of cartilage degeneration and joint inflammation, clinical patient factors, and downstream alterations in cartilage composition and morphology to provide novel insights into the pathoetiology of post-traumatic osteoarthritis (PTOA) after ACL injury and reconstruction. The study aims to enroll N=38 total patients with primary, isolated rupture to their anterior cruciate ligament (ACL), who have agreed to participate in the study and who will undergo primary surgical reconstruction by an orthopaedic physician at our two sites. Patients will undergo baseline magnetic resonance imaging (MRI), baseline clinical evaluation, and undergo a baseline blood draw. Subsequent imaging and clinical evaluations will be longitudinally performed at several postoperative timepoints up to 12 months postoperatively.

DETAILED DESCRIPTION:
Overall Study Design: This is a prospective, longitudinal cohort study of patients undergoing primary ACL reconstruction following ACL rupture. Surgical treatment and treatment timelines do not deviate from the national and international standards of care. Enrolled patients for study participation will undergo assessments involving blood, urine, and synovial fluid collection, clinical evaluation involving questionnaires and joint laxity testing, and MRI analysis.

Patient Selection and Enrollment: The participating physicians at each site will identify potential subjects from their clinics' patients according to the inclusion/exclusion criteria listed below. Based on surgical volumes at both sites, patients generally undergo ACL reconstruction 8-12 weeks after initial screening. In the preoperative timeframe, all patients will undergo standard physical therapy to address pain, swelling, and motion deficits, as is standard of care at both institutions. Arthroscopic ACL reconstruction will be performed by Dr. Bedi at the University of Michigan, by Professor Ao at Peking University, and by 5 additional surgeons at Peking University. All surgeons will utilize a standardized single-bundle technique with a hamstring or bone-patellar tendon-bone autograft.

ELIGIBILITY:
Inclusion Criteria:

* Isolated, traumatic primary anterior cruciate ligament rupture requiring surgical reconstruction
* Surgical reconstruction performed using a single-bundle technique utilizing an autograft
* No history of ipsilateral traumatic knee injury or fracture
* No evidence of Posterior Cruciate Ligament injury or more than grade 1 injury to the Medial or Lateral Collateral Ligament

Exclusion Criteria:

* Body Mass Index < 18.5 or >35 - Injury occurred longer than 4 weeks before enrollment
* Intra-articular steroid injection within 3 months of injury
* Chondral defects greater than 3 cm2 or Outerbridge grade II or higher lesions
* Pregnant women as they are not eligible for surgery

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Articular cartilage surface roughness | Baseline (preop), 12 months
  One-year change in articular cartilage surface roughness based on quantitative morphological assessment with 3D MRI.
Change in Serum Cartilage Oligomeric Matrix Protein (COMP) concentration | Baseline (preop), 12 months
  One-year change in the serum concentration of COMP, a biomarker of articular cartilage degeneration.
Change in International Knee Documentation Committee (IKDC) score | Baseline (preop), 12 months
  One year change in IKDC, a patient-reported outcome measure specific to knee injuries.

SECONDARY OUTCOMES:
Change in quantitative T2 mapping and T1rho mapping relaxation times from MRI. | Baseline (preop), 12 months
Change in concentration of biomarkers of inflammation and cartilage metabolism. | Baseline (preop), 12 months
Change in patient-reported outcome measures | Baseline (preop), 12 months
Change in knee laxity | Baseline (preop), 12 months
  Knee laxity will be measured with KT-2000 testing

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided